CLINICAL TRIAL: NCT03906344
Title: Expanded Access Use of INCB052793 to Treat a Single Patient With Myelofibrosis
Status: No longer available | Type: Expanded Access
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: I-52793-18-02
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: INCB052793

SUMMARY:
Expanded access use of INCB052793 to treat a single patient with Myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Savona, MD, Principal Investigator — Vanderbilt University Medical Center